CLINICAL TRIAL: NCT03425188
Title: Post Approval Study of the remedē System
Status: Completed | Type: Observational
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR1079
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- remedē System Subjects: Subjects who were implanted with the remedē System and actively followed as part of the remedē System Pivotal Trial at the time of study closure.

SUMMARY:
Prospective, single arm cohort study to evaluate the long-term safety, long-term effectiveness, and survival rate in subjects implanted with the remedē System.

DETAILED DESCRIPTION:
This Post Approval Study is a multi-center, prospective, single arm cohort study to evaluate the long-term safety, long-term effectiveness, and survival rate in subjects implanted with the remedē System from the remedē System Pivotal Trial. Only subjects who were implanted and actively being followed as part of the remedē System Pivotal Trial are eligible. An individual subject's participation is expected to continue to five years post remedē System implant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously implanted with the remedē System and participated in the remedē System Pivotal Trial
* In the investigator's opinion, willing and able to comply with all study requirements
* Signed Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent (including Health Insurance Portability and Accountability Act [HIPAA] authorization in the US)

Exclusion Criteria:

* There are no criteria by which a subject would be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only subjects who were implanted and actively being followed as part of the remedē System Pivotal Trial are eligible for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Germany, MD, Study Director — Respicardia, Inc.
Locations (17):
- United States (16):
  - Keck Medical Center of USC, Los Angeles, California
  - UF Health Jacksonville, Jacksonville, Florida
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Cooper Health System, Cherry Hill, New Jersey
  - Novant Clinical Research Institute Forsyth Medical Center, Winston-Salem, North Carolina
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Wesley Neurology, Cordova, Tennessee
  - Methodist Hospital, San Antonio, Texas
  - Marshfield Clinic, Marshfield, Wisconsin
- Herz-und Diabeteszentrum NRW, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 subjects enrolled in the original pivotal trial of the remede system. 94 were ongoing at the time of trial closure and therefore eligible to participate in this continuation post approval study. Pivotal trial sites with subjects ongoing at the time of study closure were invited to participate in this long-term continuation study. Subjects needed to re-consent to participate. Due to sites or subjects declining participation, not all subjects participated in this continuation study.
Groups:
- Treatment: Subjects implanted with the remedē System device, receiving active therapy and enrolled in the post approval study. This is a subset of the 151 subjects enrolled in the original pivotal trial of the remede System.
Period: Overall Study
Arm/Group | Treatment
Started | 53
Completed | 52
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Subjects implanted with the remedē System device, receiving active therapy and enrolled in the post approval study
Arm/Group | Treatment
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 50
  More than one race | 0
  Unknown or Not Reported | 1
Heart failure [Count of Participants; unit: Participants] — Defined as New York Heart Association (NYHA) Functional Class ≥ I
  Participants | 29
Apnea Hypopnea Index [Median (Inter-Quartile Range); unit: events/hour] — The number of apneas and hypopneas per hour of sleep.
  An apnea is defined by 3 characteristics:
  1. There is a drop in the peak thermal sensor excursion or alternate nasal air pressure transducer (inspiratory effort) by > 90% of baseline
  2. The duration of the event lasts at least 10 seconds
  3. At least 90% of the event's duration meets the amplitude reduction criteria for apnea
  Hypopnea defined as 30% reduction in airflow (or alternative hypopnea sensor) for ≥10 seconds over at least 90% of the event's duration that is associated with a >4% fall in oxygen saturation from baseline.
  events/hour | 41 [34 to 57]
Epworth Sleepiness Scale [Median (Inter-Quartile Range); unit: units on a scale] — The Epworth Sleepiness Scale is an assessment to measure a subject's general level of daytime sleepiness. Scores can range from 0-24, with higher scores indicating higher level of daytime sleepiness.
  units on a scale | 12 [6 to 15]

OUTCOME MEASURES:

1. Primary Outcome: 5-Year Survival Rate
Description: Assessment of survival in subjects with moderate to severe central sleep apnea being treated with the remedē System. The 5-year survival rate was estimated from Kaplan-Meier anlaysis, using time from implant to death, study exit or last contact. This analysis used all subjects enrolled in the original remede System Pivotal Trial.
Time Frame: Through 5 years
Population: All 151 subjects enrolled in the remedē System Pivotal Trial (NCT01816776) underwent an implant attempt and are included in this analysis. Longer term follow-up data from the subset of pivotal trial subjects enrolled in this post approval study was combined with the data from the pivotal trial for this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enrolled in Pivotal Trial: All subjects enrolled in the remedē System Pivotal Trial underwent an implant attempt and are included in this analysis. Subjects randomized to the Treatment group had transvenous phrenic nerve stimulation therapy activated 1 month after implant and subjects randomized to the control group had therapy activated after approximately 7 months.
Arm/Group | Enrolled in Pivotal Trial
Number analyzed (Participants) | 151
percentage of participants | 78 [71 to 85]

2. Primary Outcome: Number of Participants With Device-related Serious Adverse Events (SAEs) Through Three and Five Years
Description: Assessment of long-term safety via a summary of anticipated or unanticipated device-related SAEs. Proportion of subjects experiencing a device related SAE through the time point of interest. This analysis combined data from the original pivotal trial and this post approval study.
Time Frame: Through 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled in Pivotal Trial
Number analyzed (Participants) | 151
Participants
  3 Years | 9
  5 Years | 12

3. Primary Outcome: Number of Participants With Therapy-related Serious Adverse Events (SAEs) Through Three and Five Years
Description: Assessment of the safety of the remedē System by evaluating anticipated or unanticipated therapy-related SAEs. Proportion of subjects experiencing a therapy related SAE through the time point of interest.
Time Frame: Through 3 and 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled in Pivotal Trial
Number analyzed (Participants) | 151
Participants
  3 Years | 4
  5 Years | 4

4. Primary Outcome: Apnea-Hypopnea Index (AHI) Change From Baseline at 5 Years
Description: Change in AHI = Year 5 index - Baseline index. The Apnea-Hypopnea Index is a measurement obtained from an overnight sleep study used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The events were scored according to the 2007 "American Academy of Sleep Medicine manual for the scoring of sleep and associated events: rules, terminology and technical specifications" (Iber, et. al).
Time Frame: 5 years
Population: Includes all subjects who had 5 year sleep study results who were receiving active therapy during the sleep study. This is a subgroup of subjects from the original pivotal trial who enrolled in this post approval study and had sleep study data available at 5 years.
Measure: Median (Inter-Quartile Range); unit: Events/hour
Arm/Group | Treatment
Number analyzed (Participants) | 43
Events/hour | -22 [-42 to -7]

5. Primary Outcome: Epworth Sleepiness Scale (ESS) Change From Baseline at 5 Years
Description: Change in ESS = Year 5 score - Baseline score. The ESS is an assessment to measure a subject's general level of daytime sleepiness. Scores can range from 0-24, with higher scores indicating higher level of daytime sleepiness.
Time Frame: 5 years
Population: Includes all subjects who completed the ESS at 5 years. This is a subgroup of subjects from the original pivotal trial who enrolled in this post approval study and had data available at 5 years.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 51
units on a scale | -3 [-8 to -1]

ADVERSE EVENTS:
Time Frame: The time period includes events experienced by subjects who enrolled in this long term follow-up study, starting from time of completion of the pivotal trial and continuing through 5 years post-implant. All subjects had completed at least 2 years in the pivotal trial prior to study closure and enrollment in this long term follow-up study.
Description: In addition to the usual serious adverse event definitions, this study included any device or therapy related adverse event that required a system modification (excluding generator replacement for battery depletion within anticipated timeframe or elective explant), regardless of the procedure being to prevent one of the outcomes listed in the usual serious adverse event definitions.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 23/53
Other Adverse Events (participants affected / at risk) | 3/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=53)
HEART FAILURE (Cardiac disorders) | 3
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
HYPERTROPHIC OBSTRUCTIVE CARDIOMYOPATHY (Cardiac disorders) | 1
SINUS BRADYCARDIA (Cardiac disorders) | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
HYPOTHYROIDISM (Endocrine disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
IMPLANT SITE INFECTION (General disorders) | 1
INGROWN TOENAIL (General disorders) | 1
LEAD COMPONENT FAILURE (General disorders) | 1
LEAD DISLODGEMENT (General disorders) | 1 — The stimulation lead pulled out of the target vessel and required the lead to be replaced in order to deliver therapy
LEAD DISPLACEMENT (General disorders) | 1 — The stimulation lead remained in the target vessel but electrode position did not allow for effective therapy delivery
SIMULATION LEAD EXTRACTION (General disorders) | 1
STIMULATION LEAD PLACEMENT (General disorders) | 1
ABSCESS (Infections and infestations) | 1
APPENDICITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
WOUND INFECTION (Infections and infestations) | 1
ROTATOR CUFF TEAR (Injury, poisoning and procedural complications) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
PROSTATE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
STROKE (Nervous system disorders) | 3
PARESTHESIA (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1
URINARY TRACT PAIN (Renal and urinary disorders) | 1
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1
PAIN PUMP IMPLANT (Surgical and medical procedures) | 1
HYPERTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=53)
ATRIAL FIBRILLATION (Cardiac disorders) | 3

LIMITATIONS AND CAVEATS:
The original pivotal trial of the remede System (ClinicalTrials.gov Identifier: NCT01816776) enrolled 151 subjects and was closed following FDA approval of the PMA submission. This post approval study was initiated as a separate study to continue following as many of the 94 patients ongoing at the time of pivotal trial closure. Due to some sites declining to participate and multiple subjects declining to re-consent, the number of enrolled subjects was less than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without prior written agreement of the Sponsor, Research Institution and site Principal Investigator agree not to publish results for at least 1 year from finalization of the study database, after which time site Principal Investigator may publish or submit for publication a Manuscript without further delay subject to the sponsor having 60 days to review the proposed publication and additional 90 day provision if intellectual property is at risk to allow time for submitting patent applications.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03425188/Prot_SAP_ICF_000.pdf